CLINICAL TRIAL: NCT03981406
Title: The Impact of Palliative Care on Quality of Life, Anxiety, and Depression in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Palliative Care and Quality of Life in Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000753
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Idiopathic Pulmonary Fibrosis; Depression; Anxiety; Depressive Disorder; Anxiety Disorders; Anxiety Depression
Keywords: Palliative Care
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Depression; Anxiety Disorders; Depressive Disorder | interventions — Palliative Care; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palliative Care (Experimental): Palliative care is comprehensive, coordinated interdisciplinary care for patients and families facing a potentially life-threatening illness. This consists of specially trained teams of professionals including physicians, nurses, social workers, and chaplains that provide care and support in inpatient and outpatient settings.
  Interventions: Behavioral: Palliative Care
- Standard of Care (Placebo Comparator): Standard of care for idiopathic pulmonary fibrosis
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Palliative Care — The intervention is one visit to the Fairview Clinics and Surgery Center palliative care clinic, with follow up visits as determined by the palliative care team and the patient.
  Arms: Palliative Care
Behavioral: Standard of Care — Control group will receive standard of care treatment for IPF.
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to evaluate the effects of adding a palliative care intervention for patients with idiopathic pulmonary fibrosis (IPF) to current standard of care.

Palliative care is comprehensive, coordinated interdisciplinary care for patients and families facing a potentially life-threatening illness. This consists of specially trained teams of professionals including physicians, nurses, social workers, and chaplains that provide care and support in inpatient and outpatient settings. While the specific assistance and support provided by the Palliative Care Service depends on individual patient and family needs and preferences, it may include:

1. Pain and symptom management
2. Psychosocial and spiritual support
3. Assistance with treatment choices
4. Help in planning for care in the community

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a progressive and heterogeneous fibrotic lung disease. It is universally fatal, with an average time to death between two to five years.

Patients with IPF experience significantly diminished quality of life and increased symptom burden. Besides dyspnea, cough, fatigue, and deconditioning, patients with IPF experience significant depression and anxiety. The benefit of palliative care has been demonstrated in several other diseases, notably, in metastatic lung cancer. Patients with metastatic lung cancer who were seen by palliative care at the time of their diagnosis and throughout their disease course were found to have increased survival, improved quality of life, and received less aggressive care at the end of their life. This finding has prompted significant research in the role of palliative care in other diseases, including chronic lung disease. A non-blinded, randomized trial of a multi-disciplinary breathlessness service intervention in patients with advanced disease including cancer, chronic obstructive lung disease (COPD), interstitial lung disease (ILD), and congestive heart failure demonstrated improvement in breathlessness, anxiety, and even survival. Specific Aim 1: Determine if quality of life is improved with a palliative care intervention. Specific Aim 2: Determine if depression and anxiety symptoms are decreased with a palliative care intervention. Secondary aims include an examination of pulmonary function tests (PFT), number of hospitalizations, and overall mortality as an effect of a palliative care intervention.

ELIGIBILITY:
Inclusion Criteria:

* IPF as diagnosed by chest CT or lung biopsy, and documented by a pulmonologist in the patient's medical record
* Capacity to provide informed consent

Exclusion Criteria:

* Documented malignancy that would impact mortality within the study enrollment period
* Inability to pay for palliative care visit, insurance or personally.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline respiratory quality of life as measured by SGRQ | 6 months
  The Saint George's Respiratory Questionnaire (SGRQ) is 50-item survey with scores ranging from 0 to 100 and with higher scores indicating worse quality of life.
Change from baseline anxiety and depression symptoms as measured by HADS | 6 months
  The Hospital Depression and Anxiety Index (HADS) is a 14-item survey with scores ranging from 0 to 21 and with higher scores indicating greater depression and anxiety.
Change in prevalence of baseline depression as measured by PHQ-9 | 6 months
  The Patient Health Questionnaire (PHQ-9) is a 10-item survey with scores ranging from 1 to 27 and with higher scores indicating greater levels of depression.

SECONDARY OUTCOMES:
Change from baseline of spirometry | 6 months
  Spirometry is a commonly-used pulmonary function test (PFT) measuring lung function. Greater spirometry output will be considered a measure of greater treatment efficacy.
Change from baseline of diffusing capacity | 6 months
  Diffusing capacity is a commonly-used pulmonary function test (PFT) measuring the transfer of gas from air in the lung to the red blood cells in lung blood vessels. Greater diffusing capacity will be considered a measure of greater treatment efficacy.
Change from baseline of lung volume | 6 months
  Lung volume is a commonly-used pulmonary function test (PFT) measuring the volume of inhaled or exhaled air. Greater lung volume will be considered a measure of greater treatment efficacy.
Change from baseline of 6-minute walk distance | 6 months
  6-minute walk distance will be considered as a measure of invention efficacy, with an increase in 6-minute walk distance considered a measure of greater treatment efficacy.
Total number of hospitalizations due to any cause | 6 months
  Total number of hospitalizations due to any cause will be considered as a measure of intervention efficacy, with decrease hospitalizations in the treatment group considered a measure of greater treatment efficacy.
All-cause mortality | 6 months
  All-cause mortality will be considered as a measure of intervention efficacy, with decrease in mortality in the treatment group considered a measure of greater treatment efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Janssen K, Rosielle D, Wang Q, Kim HJ. The impact of palliative care on quality of life, anxiety, and depression in idiopathic pulmonary fibrosis: a randomized controlled pilot study. Respir Res. 2020 Jan 3;21(1):2. doi: 10.1186/s12931-019-1266-9. PMID 31900187